CLINICAL TRIAL: NCT06662422
Title: Auricular Neuromodulation and Surgical Conditions During Functional Endoscopic Sinus Surgery
Brief Title: Auricular Neuromodulation for FESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY-24-00047
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Functional Endoscopic Sinus Surgery; Vagal Nerve Stimulation; Platelet Activation
Keywords: blood loss; postoperative pain; Functional Endoscopic Sinus Surgery; Vagal Nerve Stimulation; Platelet Activation
MeSH Terms: conditions — Hemorrhage; Pain, Postoperative | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electrostimulation (Experimental): Device will be turned on to send electrostimulation.
  Interventions: Device: Spark Biomedical Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) System
- Sham - no electrostimulation (Sham Comparator): Device will be toggled to Sham so no electrostimulation will be given.
  Interventions: Device: Spark Biomedical Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) System

INTERVENTIONS:
Device: Spark Biomedical Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) System — The Spark Biomedical Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) System is a single-use electrode placed on and around the ear which provides transcutaneous auricular neurostimulation (tAN), which targets the auricular branch of the vagus nerve (ABVN) and the auriculotemporal nerve (ATN).

SUMMARY:
In this blinded prospective randomized control trial the researchers will investigate the impact of cutaneous vagal nerve stimulation on surgical conditions in patients undergoing functional and ascorbic sinus surgery (FESS). The device is an externally placed vagal nerve stimulator. The device will be applied to participants after consent and induction of anesthesia. The study team will open the randomization envelope and if the participant is assigned to stimulation the device will be turned on. In the case that the participant is assigned to the control arm, the device will be set to sham. The device will remain on for 30 minutes and removed before entering the OR. Device will be reinserted in the recovery room for another 30 minutes.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery is an important procedure for controlling a variety of sinus disease. Given the proximity to the brain and vascularity of tissues, good visualization is paramount. Intraoperative bleeding and obscure the view of the surgeon. In this study, the investigators will use a neuromodulation device that will decrease bleeding and lead to better surgical conditions during the surgery. The device used has already been studied in other bleeding environments. The investigators believe it will also work for this case. The study on Functional Endoscopic Sinus Surgery (FESS) will focus on the use of an innovative device designed to control bleeding and enhance visualization during surgery. FESS, a critical procedure for treating sinus-related conditions, often faces challenges related to bleeding and poor visibility, impacting surgical outcomes. This study aims to address these challenges by introducing a device used in other areas that promises to revolutionize the standard procedure. The device for the study, the Spark Biomedical Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) System, should decrease bleeding, a common obstacle in sinus surgery. This not only improves visibility for the surgeon but is also expected to lead to more accurate surgical interventions, reduced operation times, and fewer complications. The study will explore the efficacy and safety of this device, making a significant contribution to the field of sinus surgery and medical technology. This technology has been used in other areas, namely opiate use disorder, for which it has an FDA approval. The investigators plan to conduct a detailed investigation into the device's performance, employing a methodology that may include randomized controlled trials, adequate sample sizes, and comprehensive data collection methods. The study will assess various parameters such as the effectiveness of bleeding control, the impact on surgical duration, and overall patient outcomes. This research is not only significant for its potential to improve surgical techniques but also for its broader implications in patient care and medical innovation. By testing the hypotheses related to the device's performance and expected outcomes, the study aims to provide valuable insights that could transform the practice of sinus surgery, enhancing patient safety and surgical efficiency.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2
* Presenting for elective FESS surgery

Exclusion Criteria:

* Anti-fibrinolytic use within 30 days of enrollment
* Known or acquired coagulation disorders
* Hypercoagulable state, including morbid obesity and active smoking
* Pregnancy
* Blood transfusion with 30 days of enrollment
* History of epileptic seizures
* Presence of device such as pacemaker, cochlear prosthesis, neurostimulator
* Ear infection
* Abnormal ear anatomy which inhibits application of device
* Presence of other significant disease or disorder which under the discretion of the principal investigator could influence the results of the trial or the participant's ability to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Boezaart Score | every 15 minutes during surgical procedure
  Perioperative bleeding by Boezaart Score. Full scale is graded from Grade of 0 (clear surgical field) to 5 (severe bleeding). Higher score indicates more severe bleeding.

SECONDARY OUTCOMES:
Post-operative nausea score | during PACU stay, average PACU stay is 3 hours
  Nausea measured by presence/absence at any time during Post Anesthesia Care Unit (PACU) stay following surgical procedure
Post-operative vomiting score | during PACU stay, average PACU stay is 3 hours
  Vomiting measured by presence/absence at any time during PACU stay following surgical procedure
Visual Analog Scale (VAS) for Post-operative pain score | 30 minutes after procedure
  Pain score at initial assessment in PACU before pain medication given, once patient in alert and oriented, at approximately 30 minutes after end of surgery, measured by VAS. Full scale from 0 to 10, higher score indicates more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data and/or samples will only be used to complete this study and then they will be destroyed.

DOCUMENTS (1):
  • Informed Consent Form (2025-03-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT06662422/ICF_000.pdf